CLINICAL TRIAL: NCT04277884
Title: A Phase 3, Double-blind, Placebo-controlled, Efficacy and Safety Study of Firibastat (QGC001) Administered Orally, Twice Daily, Over 12 Weeks in Difficult-to-treat/Resistant Hypertensive Subjects
Brief Title: Firibastat in Treatment-resistant Hypertension
Acronym: FRESH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Quantum Genomics SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QGC001-3QG1
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — firibastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Firibastat (Experimental): Capsules
  Interventions: Drug: Firibastat
- Placebo (Placebo Comparator): Matching capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Firibastat — Oral administration 2×250 mg capsules bid
  Other Names: QGC001
  Arms: Firibastat
Drug: Placebo — Oral administration 2 capsules bid
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, multicenter, efficacy and safety study of firibastat (QGC001) administered po bid over 12 weeks in male and female subjects ≥18 years of age at Screening, with uncontrolled primary HTN. Subjects will be randomized 1:1 to investigational product (IP) and will receive either firibastat (QGC001) or matching placebo on top of their current chronic antihypertensive treatments.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effects of administration of firibastat (QGC001) 500 mg oral (po) twice daily (bis in die [bid]) on blood pressure (BP) over 12 weeks in subjects with uncontrolled primary HTN.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age at Screening
* Diagnosis of primary HTN for at least 6 months prior to Screening

Exclusion Criteria:

* Known or suspected secondary HTN (eg, hyperaldosteronism, renovascular HTN, pheochromocytoma, Cushing's disease).
* Automated office SBP >180 mmHg or DBP >110 mmHg at the Screening or Inclusion Visit (Visit 2, Day 1) and confirmed by a second measurement within 30 minutes to 1 hour.
* Known hypertensive retinopathy (Keith-Wagener Grade 3 or Grade 4) and/or hypertensive encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure at office (mmHg) | From Day 1 to Day 84
  Automatic Office Blood Pressure measurement

SECONDARY OUTCOMES:
Diastolic Blood Pressure at office (mmHg) | From Day 1 to Day 84
  Automatic Office Blood Pressure measurement
Mean 24-hour ambulatory Systolic Blood Pressure (mmHg) | From Day 1 to Day 84
  Ambulatory Blood Pressure Monitoring
Mean 24-hour ambulatory Diastolic Blood Pressure (mmHg) | From Day 1 to Day 84
  Ambulatory Blood Pressure Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: George Bakris, MD, Principal Investigator — AHA Comprehensive Hypertension Center
Locations (20):
- United States (15):
  - Central Alabama Research, Birmingham, Alabama
  - Marvel Clinical Research, Huntington Beach, California
  - Orange County Research Center, Tustin, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Apex Medical Research, Chicago, Illinois
  - Cedar Crosse Research Center, Chicago, Illinois
  - ClinEdge - Chear Center, The Bronx, New York
  - Sterling Research Group - Cincinnati / Mount Auburn, Cincinnati, Ohio
  - Insearch - Punzi Medical Center, Carrollton, Texas
  - ClinEdge - Dayton Clinical Research, Dayton, Texas
  - Juno Research - Corporate Office, Houston, Texas
  - Insearch - R&H Clinical Research, Katy, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
- Fakultní nemocnice v Motole, Prague, Czechia
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, Grand Est, France
- Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Germany
- Ambulatorium Barbara Bazela, Elblag, Żuławy, Poland
- Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khosla J, Aronow WS, Frishman WH. Firibastat: An Oral First-in-Class Brain Aminopeptidase A Inhibitor for Systemic Hypertension. Cardiol Rev. 2022 Jan-Feb 01;30(1):50-55. doi: 10.1097/CRD.0000000000000360. PMID 33027067